CLINICAL TRIAL: NCT01731782
Title: Evaluation of a TAP Block as Part of an Enhanced Recovery Pathway in Laparoscopic Colorectal Surgery: A Prospective, Randomized, Double-blinded Multi-institution Trial
Brief Title: Evaluation of a TAP Block Given During Laparoscopic Colorectal Surgery to Help Control Pain
Acronym: TAP Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 02-12-03
Record Dates: First submitted 2012-10-19; First posted 2012-11-22 (Estimated); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Disease
Keywords: colorectal surgery
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bupivacaine (Active Comparator): bupivacaine-0.5ml/kg of 25% bupivacaine for maximum of 30ml
  Interventions: Drug: bupivacaine
- normal saline (Placebo Comparator): Normal saline placebo-0.5ml/kg of 0.9% normal saline (max of 30ml)to mimic bupivacaine
  Interventions: Drug: normal saline placebo (for bupivacaine)

INTERVENTIONS:
Drug: bupivacaine
  Other Names: Marcaine
  Arms: bupivacaine
Drug: normal saline placebo (for bupivacaine) — Normal saline to mimic bupivacaine
  Arms: normal saline

SUMMARY:
Patients experience pain after surgery mostly from their abdominal wounds, even when those wounds are small. Decreasing that pain has many benefits. It improves comfort, decreases stress response and might improve the outcome of the surgery. Local anesthesia (which is a numbing agent given directly at the site of pain via a needle) is given to decrease the pain that is felt after surgery and decrease the need for strong pain medications which can have negative side effects.

One promising way to give local pain medication is called the "transversus abdominis plane" or TAP block. This method works by directly blocking the nerves in the abdomen that are the cause of the pain patients feel in their incision after surgery. This is done by injecting a numbing agent (Bupivacaine) into the area of their abdomen where their nerves are located that cause pain.

In the case of nerves that carry sensation, bupivacaine blocks the pain sensation traveling in a particular nerve.

Patients will be randomized (like a flip of a coin) to receive either a normal saline injection or the bupivacaine injection.

The purpose of this study will be to prove the effectiveness of local anesthetic given via a TAP block in improving postoperative pain, decreasing the use of pain medications, decreasing postoperative nausea and vomiting and improve surgical outcomes such as hospital length of stay in laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
Using standard surgical procedures, the surgeon will proceed with the planned laparoscopic surgery. All procedures will be done by straight laparoscopic technique according to standard of care. At the completion of the procedure, and under laparoscopic control, patients will have a TAP block placed by the attending surgeon. The clinical research nurse involved in the research will prep the solution to be injected and the surgeon will be blinded as to whether the patient will be receiving normal saline or Marcaine in the TAP blocks. The block will be administered between the costal margin and iliac crest in the anterior axillary line. A Braun Stimuplex A insulated needle (80 mm 21 gauge) with 0.5 mL/kg solution (max of 30 ml) is passed through the skin, and then continued until two distinct "pops" are felt, which indicates the needle piercing each of the two fascial layers. The needle is then deemed to be in the inter-muscular plane between internal oblique and transversus abdominis muscles respectively, to target the spinal nerves in this plane. The laparoscope will be visualizing for the needle tip to ensure that it does not penetrate the peritoneum or inject pre-peritoneally. The local anesthetic is infiltrated in two separate injections into the same plane on each side. If a sub-peritoneal bleb is seen to be raised by the laparoscope, then the needle will be withdrawn slightly. Two thirds of the solution is injected, and the needle is withdrawn 5 mm and the remaining solution is injected. If injecting in the correct plane, then a smooth raised area of fluid, covered by transversus will be seen via the laparoscope. This procedure is repeated on the patients other side, to complete a bilateral block. Depending on their randomization, patients will receive one of the following solutions:

Group A: Represents the control group and will receive 0.5 ml/kg of 0.9% normal saline for a maximum of 30 ml.

Group B: Represents the experimental group and will receive 0.5 ml/kg of 0.25% Marcaine (bupivacaine) for a maximum of 30 ml.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have benign or malignant colonic or rectal disease that are being scheduled for laparoscopic colorectal resection.
2. Subjects who are 18 years of age and older
3. Subjects of either sex
4. Subjects who are willing and able to adhere to protocol requirements, agree to participate in the study program and provide written and informed consent.

Exclusion Criteria:

1. Subjects who undergo conversion to the open approach will be excluded from the analysis, as the block will be given at the end of the procedure and is being evaluated for laparoscopic cases.
2. Subjects who are pregnant.
3. Subjects with a medical condition that may interfere with the use of the study medication Bupivicaine.
4. Subjects who have another condition or general disability or infirmity that in the opinion of the investigator precludes further participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Conor P Delaney, MD.,PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine: bupivacaine-0.5ml/kg of 25% bupivacaine for maximum of 30ml
  bupivacaine
Period: Overall Study
Arm/Group | Bupivacaine | Normal Saline
Started | 41 | 38
Completed | 41 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Normal Saline | Total
Number analyzed (Participants) | 41 | 38 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.34 (14.16) | 64.82 (13.11) | 66.12 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain as Measured by Pain Score
Description: Pain measured via score of 1 to 5, with 1 being no pain and 5 being the worst pain
Time Frame: up to 10 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine | Normal Saline
Number analyzed (Participants) | 41 | 38
score on a scale | 2.60 (2.09) | 3.46 (1.92)

2. Secondary Outcome: Percent of Analgesics Used as Measured by Patient Report
Time Frame: Up to 30 days after surgery
Measure: Mean (Standard Deviation); unit: percentage of analgesics used
Arm/Group | Bupivacaine | Normal Saline
Number analyzed (Participants) | 41 | 38
percentage of analgesics used | 0.80 (0.52) | 1.79 (0.72)

3. Other Pre Specified Outcome: Number of Nausea/Vomiting Episodes
Time Frame: up to 10 days
Measure: Number; unit: Episodes
Arm/Group | Bupivacaine | Normal Saline
Number analyzed (Participants) | 41 | 38
Episodes | 10 | 9

4. Other Pre Specified Outcome: Length of Hospital Stay
Time Frame: up to 10 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bupivacaine | Normal Saline
Number analyzed (Participants) | 41 | 38
days | 3.15 (2.03) | 2.87 (1.58)

5. Other Pre Specified Outcome: Day of Return of Bowel Function
Description: Log the day bowel function returns by day postoperative that flatus returns and has first stool
Time Frame: daily after surgery until discharge up to 10 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 30 days postop
Arm/Group | Bupivacaine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/38
Other Adverse Events (participants affected / at risk) | 0/41 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine (N=41) | Normal Saline (N=38)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — Patient remained in the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT01731782/Prot_SAP_000.pdf